CLINICAL TRIAL: NCT05686967
Title: MitoQ Supplementation for Restoring Aerobic Exercise Training Effects on Endothelial Function in Postmenopausal Women
Brief Title: MitoQ and Exercise Effects on Vascular Health
Acronym: MITO-STEP
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 22-1521; R56AG072094 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2023-01-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aging; Menopause
Keywords: vascular health; exercise; oxidative stress
MeSH Terms: conditions — Motor Activity | interventions — mitoquinone; mitoquinol; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and assessor will be blinded to MitoQ or Placebo. Participants will not be blinded to exercise or no exercise; investigators and assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise plus MitoQ (Experimental): Moderate intensity aerobic exercise, 50 minutes of treadmill exercise, 65-75% of maximal heart rate, 3 d/week for 10 weeks plus experimental MitoQ, 20mg/d.
  Each MitoQ capsule contains 20 mg of mitoquinol mesylate. Dosage: 20 mg orally per day for 10 weeks.
  Interventions: Dietary Supplement: MitoQ; Behavioral: Aerobic exercise
- Aerobic Exercise plus Placebo (Placebo Comparator): Moderate intensity aerobic exercise, 50 minutes of treadmill exercise, 65-75% of maximal heart rate, 3 d/week for 10 weeks plus matching placebo capsule/d for 10 weeks.
  Matched placebo capsules.
  Interventions: Dietary Supplement: Placebo; Behavioral: Aerobic exercise
- No Exercise plus MitoQ (Experimental): No exercise plus experimental MitoQ, 20mg/d. Each MitoQ capsule contains 20 mg of mitoquinol mesylate. Dosage: 20 mg orally per day for 10 weeks.
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ is a biochemically modified form of ubiquinol
  Other Names: Mitoquinol
  Arms: Aerobic Exercise plus MitoQ; No Exercise plus MitoQ
Dietary Supplement: Placebo — Each placebo capsule contains inert excipient and is identical in appearance
  Arms: Aerobic Exercise plus Placebo
Behavioral: Aerobic exercise — Moderate intensity aerobic exercise on the treadmill
  Arms: Aerobic Exercise plus MitoQ; Aerobic Exercise plus Placebo

SUMMARY:
An impairment in vascular function can lead to the development of age-associated cardiovascular disease (CVD), the leading cause of death in postmenopausal women. Regular aerobic exercise (AE) benefits vascular function in older men by reducing oxidative stress, however, similar AE training improvements are diminished or absent in postmenopausal women. not using estrogen-based hormone therapy. Vascular function and oxidative stress are improved with AE training in postmenopausal women treated with E2, suggesting an essential role of E2 in vascular adaptations to AE in women. Clinical use of E2 is contraindicated for this purpose, thus establishing alternative pharmacological approaches that could be administered as a substitute for E2 to improve AE signaling for vascular benefits and reducing CVD risk in E2-deficient postmenopausal women is biomedically important. The mitochondrial-targeted antioxidant MitoQ may be an alternative to E2 for restoring AE benefits in E2-deficient postmenopausal women given its recently established effectiveness for reducing oxidative stress and improving vascular function in that population. Accordingly, the overall aim of this application is to assess the efficacy of a 12-week randomized controlled trial of moderate intensity AE training combined with oral MitoQ (20 mg/d) compared to AE+oral placebo (PL) or No AE+MitoQ on vascular vasodilatory function (brachial artery flow-mediated dilation; FMD) in healthy E2-deficient postmenopausal women. Insight into the causes for the improvement related to molecules (e.g., nitric oxide) that promote vasodilation, mitochondrial function, oxidative stress, and the influence of "circulating factors" will also be obtained. We hypothesize that AE+MitoQ will improve both FMD > AE+PL and > No AE+MitoQ, and that No AE+MitoQ will improve FMD > AE+PL. The greater improvements in endothelial function with AE+MitoQ vs. both AE+PL and No AE+MitoQ, and with No AE+MitoQ vs. AE+PL will be mediated by greater improvements in nitric oxide production, mitochondrial function, and mitochondrial and oxidative stress linked, at least in part, to changes in "circulating factors". The expected results from this study will establish the efficacy of MitoQ for restoring AE-vascular signaling in E2-deficient postmenopausal women and will provide the foundation for development of evidence-based guidelines for sex-specific AE programs for improving vascular health and preventing CVD in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* resting blood pressure <140/90 mmHg;
* fasted glucose <126 mg/dL;
* sedentary/recreationally active (<2 days/wk vigorous exercise);
* healthy, as determined by medical history, physical examination, standard blood chemistries (chemistry panel, CBC and circulating thyroid levels) and ECG at rest and during exercise;
* nonsmokers;
* no use of medications that might influence cardiovascular function (i.e., antihypertensive, lipid lowering medications, blood thinners);
* no use of vitamin supplements or anti-inflammatory medications, or willing to stop 1 month prior to enrollment and for the duration of the study;
* no use of HT for at least 6 months;
* body mass index <40kg/m2.

Exclusion Criteria:

* Volunteers will be excluded from the study if they have contraindications to MitoQ or AE.
* acute liver disease, history of venous thromboembolic events, preexisting or active cardiac, renal or hepatic disease, history of stomach ulcer or bleeding or epilepsy or other seizure disorder;
* diabetes, active infection, disease that affects the nervous system,
* an abnormal resting ECG, angina and/or ECG evidence of acute myocardial ischemia during the exercise test (development of ST-segment depression of more than 0.3 mV that is either horizontal, down-sloping, or slowly upsloping -less than 1 mvolt/sec and lasts more than 0.08 sec; ST elevation; chest pain or discomfort), bundle branch blocks, A-V block greater than first degree, arrhythmias;
* chronic infections;
* thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement;
* orthopedic or other problems that would interfere with participation in the exercise program

The volunteers who choose to participate will do so with the understanding that they will be randomly assigned to study groups that involve either AE+PL (33% chance), No AE+MitoQ (33% chance) or AE+MitoQ (33% chance).

Ages: 50 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 22 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Endothelial function at 10 weeks | Baseline and after 10 weeks
  Brachial artery flow-mediated dilation

OTHER OUTCOMES:
Change from baseline in Change in Suppression of endothelial function by mitochondrial oxidative stress at 10 weeks | Baseline and 10 weeks
  Change in brachial artery flow-mediated dilation with acute supratherapeutic MitoQ dosed at 160mg
Change from baseline in Serum exposure-induced endothelial cell reactive oxygen species production at 10 weeks | Baseline and 10 weeks
  Endothelial cell whole-cell (CellROX) and mitochondria-specific (MitoSOX) reactive oxygen species levels after treatment with serum from subjects
Change from baseline Serum exposure-induced endothelial cell nitric oxide production from at 10 weeks | Baseline and 10 weeks
  Endothelial cell DAF-FM before and after addition of 200 µM Ach will quantify the capacity of HUVECs to generate nitric oxide after treatment with serum from subjects

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie L Moreau, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Center, Clinical Translational Research Center and Exercise Research Laboratory, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No